CLINICAL TRIAL: NCT02768922
Title: Aphasia Telerehabilitation Post Stroke
Brief Title: Aphasia Telerehabilitation
Acronym: AT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnaas Rehabilitation Hospital (Other)
Collaborators: South-Eastern Norway Regional Health Authority (Other)
Responsible Party: Principal Investigator, Frank Becker, Clinical Medical Director, Associate professor, Sunnaas Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21524505
Record Dates: First submitted 2016-04-25; First posted 2016-05-11 (Estimated); Last update posted 2019-04-01 (Actual); Status verified 2019-03

CONDITIONS: Stroke; Aphasia
Keywords: Telemedicine; Telerehabilitation; Speech and language therapy
MeSH Terms: conditions — Stroke; Aphasia; Communication Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aphasia telerehabilitation (Experimental): Speech and language therapy is given by telemedicine to improve expressive language function. The therapy will include knowledge based tasks of aphasia rehabilitation including training of language forms and overall functional communication. A special emphasis will be put on naming training. The telerehabilitation will be given in a addition to standard face-to-face aphasia rehabilitation
  Interventions: Other: Aphasia telerehabilitation; Other: Standard face-to-face aphasia rehabilitation
- Control (Active Comparator): Control Group receives standard face-to-face aphasia rehabilitation
  Interventions: Other: Standard face-to-face aphasia rehabilitation

INTERVENTIONS:
Other: Aphasia telerehabilitation — Speech and language therapy delivered by speech-language pathologist via computer and telemedicine
  Arms: Aphasia telerehabilitation
Other: Standard face-to-face aphasia rehabilitation — Speech and language therapy delivered by speech-language pathologist face-to-face (treatment as usual)

SUMMARY:
This study aims at contributing with scientific evidence to the field of aphasia telerehabilitation. In Norway today, there is an unmet need for language training in post stroke aphasia and not all patients are offered language training. Early start of aphasia rehabilitation and satisfying intensity do not seem to be standard clinical practice. Language training by telemedicine could improve this situation, and this study seeks to answer the question whether aphasia rehabilitation delivered by videoconference can improve language function in aphasia post stroke.

DETAILED DESCRIPTION:
BACKGROUND:

About 25 % of all stroke cases lead to aphasia. Aphasia can include difficulties with speech production and comprehension, as well as reading and writing impairment. Language impairment affects post stroke rehabilitation in a negative manner. Quality of life is reduced in persons with aphasia compared to stroke victims without aphasia. Speech and language therapy is the main form of aphasia rehabilitation. The most updated Cochrane review indicates that intensive speech and language therapy is more effective than therapy of lower intensity. Current aphasia services in Norway do not seem to be in accordance with the national guidelines for treatment and rehabilitation of stroke. The capacity for aphasia rehabilitation at the community level is too small and there is a lack of speech -language pathologists (SLPs). Language training by videoconference could improve this unmet need for language training in post stroke aphasia. The literature within this field is however sparse and there is a substantial lack of studies showing the effectiveness of telerehabilitation. Financed by the Norwegian Foundation for Health and Rehabilitation, the investigators have earlier performed a feasibility study at Sunnaas Rehabilitation Hospital in cooperation with the Norwegian Centre for Integrated Care and Telemedicine. This feasibility study showed that language training by videoconference is feasible with regard to technical, practical and rehabilitation aspects. The feasibility study laid ground for a larger and controlled study.

OBJECTIVE:

The project aims at contributing with scientific evidence to the field of aphasia telerehabilitation. The objective of this randomized controlled clinical trial is to investigate the feasibility and effectiveness of speech and language training given by videoconference.

DESIGN:

The study will be conducted as a pragmatic exploratory randomized controlled clinical trial (RCT) with an intervention and a control group. The patients will be assessed at inclusion and before randomization (baseline), and at 4 weeks and 4 months post randomization. Testing is blinded.

PARTICIPANTS:

Patients will be recruited from the stroke units at Oslo University Hospital, Akershus University Hospital, Østfold Hospital,and Bærum Hospital. Patients, who are admitted for rehabilitation at Sunnaas Rehabilitation Hospital, will also be included. In addition, patients earlier treated or on the waiting list at Sunnaas Rehabilitation Hospital, will be invited to participate. The investigators will also try to recruit patients from other rehabilitation institutions, and in cooperation with SLPs in the region of Oslo, Østfold and Akershus. The investigators will also invite for participation through the Aphasia Association of Norway (user organization).

The study aims at including 40 participants in each group, with a total number of 80 subjects. The investigators will include patients with aphasia in all stages following stroke including naming impairment. Patients under the age of 16 years and patients, who are unable to perform five hours of speech and language therapy per week due to medical or cognitive reasons, will be excluded.

INTERVENTION:

The intervention group will receive speech and language therapy via videoconference while the control group will not receive any specific therapy as part of this study. Both groups will receive standard aphasia rehabilitation (usual care). The amount of standard aphasia rehabilitation (usual care) will be logged in all participants. Participants in the intervention group will receive speech-language training (SLT) for five hours a week over four consecutive weeks. The SLT will be performed by an SLP using videoconference via internet from Sunnaas Rehabilitation Hospital to the laptop in the patient's home, or rehabilitation/nursing ward. To secure treatment fidelity and replication for future studies, the investigators have used the template for intervention description and replication (TiDieR) checklist and guide to describe the intervention. The investigators will use the technical solution "Cisco Jabber Video/Acano" and the remote control software "LogMeIn", in the telerehabilitation that is given.

PROCEDURES:

The stroke units will inform potential participants about the project and refer them to Sunnaas Rehabilitation Hospital for further investigation. Potential participants, who are patients at Sunnaas Rehabilitation Hospital, receive information about the project and an invitation to take part in the trial. For recruitment from other rehabilitation institutions, local speech and language therapists, and for members of the Aphasia association of Norway, advertising in form of a flyer and a brochure is used. After referral an ambulatory visit by the PhD-fellow or research SLP will be performed. Detailed information about the project will be provided and the research investigator will request an informed consent before carrying out baseline testing. Baseline assessment is blinded as it is performed before group allocation. The four weeks control and follow-up-testing is performed by external SLPs blinded to group allocation. Directly after the intervention period (four weeks), the participant will be visited at home or come to the outpatient clinic at Sunnaas Rehabilitation Hospital. The laptop will be retrieved and assessment performed. The control group will be tested at the corresponding time point. A further follow-up assessment will be performed four months post randomization in all participants. The four weeks control and follow-up-testing is performed by external SLPs blinded to group allocation.

OUTCOME MEASURES:

To investigate the effect of aphasia rehabilitation delivered by telemedicine, the investigators have chosen to look especially on naming as a measure of expressive language function. The investigators want to regard the prolonged effect of aphasia telerehabilitation on language function. Further on the investigators want to see the effect immediately after intervention and on other language functions than naming. The investigators also want to investigate whether SLT by videoconference can affect quality of life, if it is feasible and how persons with aphasia and therapists experience the telerehabilitation.

For the assessment of language functioning, the Norwegian Basic Aphasia Assessment (NGA) with the subtests conversational interview, naming, repetition and comprehension will be used.To assess the ability of sentence production, the investigators will use the Verb and Sentence Test (VAST) subtest sentence production. Functional communication will be assessed using Communicative Effectiveness Index (CETI). Quality of life will be assessed using Stroke and Aphasia Quality of Life scale (SAQOL-39). In addition, the experiences of patients, relatives and therapists with the telerehabilitation services will be assessed using a questionnaire as well as semi-structured interviews with selected patients. There will be an interview with the SLPs performing the telerehabilitation.

Primary endpoint: Naming ability four months post randomization.

Secondary endpoints:

* Language functions other than naming (repetition, comprehension, sentence production) four months post randomization.
* Functional communication and quality of life four months post randomization..
* Naming and other language functions immediately after intervention.
* How the telerehabilitation is experienced by patients and SLPs.
* Feasibility of telerehabilitation with regards to ethical, technical, logistic, patient and data safety aspects.

ANALYSES AND STATISTICS:

The investigators will use an intention to-treat (ITT) analysis. The trial is a longitudinal study that will give continuous repeated measurements, and the data will be analyzed using Mixed-models. Data will be examined for differences over time and between groups. Subgroup analysis will be performed to explore factors considered to affect the outcome of the trial like differences in time since onset of stroke or demographic and stroke-related factors. Qualitative data collected from semi-structured interviews will be suitably coded.

ELIGIBILITY:
Inclusion Criteria:

* Patients with aphasia following stroke (all stages of aphasia post stroke)
* Aphasia including naming impairment (percentile score of 70 or lower on the NGA - subtest naming)

Exclusion Criteria:

* Age: < 16 years
* Patients who are unable to perform 5 hours of speech and language therapy per week due to medical or cognitive reasons (Including vision and hearing impairment)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2016-05-03 (Actual); Primary Completion 2018-09-27 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Naming ability assessed by NGA | four month post randomization
  Will be assessed by the Norwegian Basic Aphasia Assessment (NGA) subtest "naming"

SECONDARY OUTCOMES:
Language function other than naming (repetition) assessed by NGA | four month post randomization
  Repetition will be assessment by the Norwegian Basic Aphasia Assessment (NGA) subtest "repetition".
Language function other than naming (comprehension ) assessed by NGA | four month post randomization
  Comprehension will be assessment by the Norwegian Basic Aphasia Assessment (NGA) subtest "comprehension".
Sentence Production by VAST | four month post randomization
  Sentence production will be assessed by the Verb and sentence test (VAST)
Sentence Production by VAST | immediately after intervention (4 weeks)
  Sentence production will be assessed by the Verb and sentence test (VAST)
Functional communication assessed by CETI | four month post randomization
  Functional communication will be assessed using Communicative Effectiveness Index (CETI).
Naming immediately after intervention assessed by NGA | immediately after intervention (4 weeks)
  Assessed by Norwegian Basic Aphasia Assessment (NGA) subtest "naming"
Repetition immediately after intervention assessed by NGA | immediately after intervention (4 weeks)
  Assessed by Norwegian Basic Aphasia Assessment (NGA) subtest "repetition"
Comprehension immediately after intervention assessed by NGA | immediately after intervention (4 weeks)
  Assessed by Norwegian Basic Aphasia Assessment (NGA) subtest "comprehension"
Experiences of patients with the telerehabilitation by questionnaire | four month post randomization
  Will be assessed by a questionnaire
Experiences of patients with the telerehabilitation by semi-structured interviews. | through study completion, an average of 2 year
  Will be assessed by semi-structured interviews with selected patients
Experiences of SLPs with the telerehabilitation by semi-structured interviews | through study completion, an average of 2 year
  Will be assessed by semi-structured interviews with selected patients
Quality of life assessed by SAQOL-39. | four month post randomization
  Quality of life will be assessed using Stroke and Aphasia Quality of Life scale (SAQOL-39).

CONTACTS AND LOCATIONS:
Overall Officials: Frank Becker, PhD, Study Director — Sunnaas Rehabilitation Hospital
Locations (1):
- Sunnaas Rehabilitation Hospital, Nesoddtangen, Norway

IPD SHARING:
Plan to Share IPD: Yes
The project will result in a Doctor of Philosophy (PhD) -thesis based on articles in international peer-reviewed scientific journals. In addition, the results of the project will be disseminated through national and international conference contributions as well as Norwegian publications in scientific journals, journals of user organizations and media contributions.

REFERENCES:
- [Derived] Ora HP, Kirmess M, Brady MC, Sorli H, Becker F. Technical Features, Feasibility, and Acceptability of Augmented Telerehabilitation in Post-stroke Aphasia-Experiences From a Randomized Controlled Trial. Front Neurol. 2020 Jul 31;11:671. doi: 10.3389/fneur.2020.00671. eCollection 2020. PMID 32849176
- [Derived] Ora HP, Kirmess M, Brady MC, Winsnes IE, Hansen SM, Becker F. Telerehabilitation for aphasia - protocol of a pragmatic, exploratory, pilot randomized controlled trial. Trials. 2018 Apr 2;19(1):208. doi: 10.1186/s13063-018-2588-5. PMID 29606148
- See also: pdf-file of Norwegian publication presenting the pilot study that led to this RCT — http://norsklogopedlag.no/Userfiles/Upload/Files/4-13_språktrening.pdf
- See also: pdf-file of full report from the pilot study (Norwegian) — https://www.extrastiftelsen.no/prosjekter/spraktrening-rett-hjem/